CLINICAL TRIAL: NCT07069140
Title: Effectiveness of an Oral Care Protocol Based on Lactoferrin Toothpaste and Mouthwash in Pregnant Women for the Prevention of Periodontal Disease: A Randomized Controlled Clinical Trial
Brief Title: Lactoferrin-Based Oral Care for Periodontal Health in Pregnancy
Acronym: LBC-PREG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LBCGEST
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Periodontal Disease; Gingivitis; Oral Microbiota
Keywords: Lactoferrin; Pregnancy; Periodontal Disease; Oral Microbiota; Dental Plaque; Gingivitis; Non-surgical Periodontal Therapy; Toothpaste; Mouthwash; LBC Complex; Maternal Oral Health; Randomized Controlled Trial; Oral Hygiene in Pregnancy
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Dental Plaque | interventions — Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin Toothpaste + Mouthwash (Experimental): Participants randomized to this arm will undergo professional dental hygiene sessions every 3 months and will perform home oral care using both a lactoferrin-based toothpaste and a lactoferrin-based mouthwash (Emoform Glic). They will be instructed to brush their teeth twice daily using the toothpaste and to rinse with 10 mL of mouthwash for 60 seconds twice daily, for a total study duration of 6 months. The intervention aims to evaluate the added benefit of combining both products on plaque accumulation and periodontal inflammation in pregnant women between the 4th and 8th month of gestation.
  Interventions: Drug: Lactoferrin-based Toothpaste and Mouthwash (Emoform Glic)
- Lactoferrin Toothpaste (Active Comparator): Participants randomized to this arm will also undergo professional dental hygiene sessions every 3 months. For home care, they will use only the lactoferrin-based toothpaste (Emoform Glic), brushing twice daily for 2 minutes following standard oral hygiene instructions. No mouthwash will be used. This group serves as the active comparator to determine whether the addition of the lactoferrin-based mouthwash provides any significant clinical advantage.
  Interventions: Drug: Lactoferrin-Based Toothpaste Only (Emoform Glic)

INTERVENTIONS:
Drug: Lactoferrin-based Toothpaste and Mouthwash (Emoform Glic) — Participants in the experimental arm will receive professional supragingival and subgingival dental hygiene sessions every three months over a six-month period. In addition, they will follow a home oral care protocol consisting of twice-daily use of a lactoferrin-based toothpaste and a lactoferrin-based mouthwash, both commercially available as Emoform Glic (Polifarma Benessere S.r.l.). The toothpaste will be applied with a soft-bristle toothbrush for two minutes, and the mouthwash will be used at a dosage of 10 mL, rinsed for 60 seconds after toothbrushing, twice a day. The intervention aims to assess whether the combined use of lactoferrin-based toothpaste and mouthwash can enhance clinical outcomes related to plaque accumulation and periodontal inflammation in pregnant women between the fourth and eighth month of gestation.
  Arms: Lactoferrin Toothpaste + Mouthwash
Drug: Lactoferrin-Based Toothpaste Only (Emoform Glic) — Participants in the control arm will also undergo professional dental hygiene sessions every three months for a total duration of six months. At home, they will follow an oral hygiene protocol limited to the twice-daily use of a lactoferrin-based toothpaste (Emoform Glic, Polifarma Benessere S.r.l.), applied with a soft-bristle toothbrush for two minutes. No mouthwash will be used in this arm. The purpose of this intervention is to evaluate the effectiveness of lactoferrin toothpaste alone and to serve as an active comparator for assessing the additional benefit of the mouthwash in improving periodontal parameters.
  Arms: Lactoferrin Toothpaste

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of a lactoferrin-based oral hygiene protocol in improving periodontal health during pregnancy. Forty pregnant women between the fourth and eighth month of gestation will be enrolled and randomly assigned to one of two groups. The trial group will undergo professional dental cleaning every three months and will perform home oral hygiene using both a lactoferrin-based toothpaste and a lactoferrin-based mouthwash (Emoform Glic) twice daily. The control group will follow the same schedule of professional dental cleanings but will use only the lactoferrin-based toothpaste (Emoform Glic) at home. The primary objective is to assess the reduction in dental plaque, measured by the Plaque Index (PI). Secondary outcomes include improvements in gingival inflammation, probing pocket depth, clinical attachment level, and other periodontal indices. Participants will be followed for six months, with evaluations conducted at baseline, 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged between 18 and 45 years
* Gestational age between 14 and 28 weeks at the time of enrollment (second trimester)
* Diagnosis of periodontitis according to the 2017 World Workshop classification (Stages I-III, Grades A-B)
* Presence of at least 20 natural teeth
* Willingness to comply with study procedures and attend follow-up visits
* Signed informed consent

Exclusion Criteria:

* History of systemic diseases that could affect periodontal status (e.g., diabetes mellitus, immunosuppression)
* Antibiotic or anti-inflammatory therapy within 3 months prior to enrollment Current use of probiotics, antioxidant supplements, or medicated mouthwashes
* Periodontal treatment within 6 months before enrollment
* High-risk pregnancy or pregnancy complications (e.g., preeclampsia, gestational diabetes)
* Smoking or tobacco use
* Known allergy to any of the investigational product components
* Participation in another clinical trial within the previous 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-identified females only. Participants must be biologically female and currently pregnant at the time of enrollment.
Enrollment: 40 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in dental plaque accumulation measured by Plaque Index (PI) | Baseline (T0) to Month 6 (T3)
  The primary outcome of this study is the change in dental plaque levels assessed using the Plaque Index (PI) developed by Silness and Löe. This index measures the thickness of dental plaque at the gingival margin. For each participant, four surfaces of each tooth (buccal, lingual, mesial, and distal) are examined and scored on a scale from 0 to 3. A score of 0 corresponds to the absence of plaque. A score of 1 indicates the presence of a plaque film only visible with a disclosing agent or by using a periodontal probe. A score of 2 indicates visible moderate plaque accumulation at the gingival margin, while a score of 3 reflects heavy plaque deposits within the gingival sulcus and around the gingival margin. The final PI for each subject is obtained by calculating the mean of all recorded surface scores. This measure provides a continuous variable where higher scores represent greater plaque accumulation and worse oral hygiene. The index will be recorded at four time points: baseline (

SECONDARY OUTCOMES:
Change in gingival bleeding measured by Bleeding on Probing (BoP) | Baseline (T0) to Month 6 (T3)
  This outcome assesses the degree of gingival inflammation by measuring the percentage of sites exhibiting bleeding after gentle probing of the gingival sulcus using a calibrated periodontal probe. BoP is recorded dichotomously, assigning a score of 0 to non-bleeding sites and 1 to bleeding sites. The final BoP score is calculated as the proportion of bleeding sites over the total number of examined sites, expressed as a percentage. Higher percentages indicate more severe inflammation. BoP values will be collected at baseline and at 1, 3, and 6 months to compare the anti-inflammatory effectiveness of the two home care protocols.
Change in periodontal pocket depth measured by Probing Pocket Depth (PPD) | Baseline (T0) to Month 6 (T3)
  This outcome measures the depth of the gingival sulcus or periodontal pocket using a periodontal probe. Probing Pocket Depth (PPD) is defined as the distance, in millimeters, from the free gingival margin to the bottom of the sulcus or pocket. Six sites per tooth are examined, and the average depth per participant is calculated. Deeper pockets reflect more severe periodontal involvement. PPD scores will be compared between the experimental and control groups at baseline, 1, 3, and 6 months to evaluate the effect of the lactoferrin-based mouthwash in addition to toothpaste.
Change in connective tissue attachment loss measured by Clinical Attachment Level (CAL) | Baseline (T0) to Month 6 (T3)
  Clinical Attachment Level (CAL) represents the cumulative loss of periodontal supporting tissue and is calculated as the distance from the cementoenamel junction (CEJ) to the base of the sulcus or periodontal pocket. It is measured in millimeters at six sites per tooth using a calibrated probe. Improvements in CAL over time reflect periodontal healing or stabilization.
Change in gingival inflammation severity measured by Modified Gingival Index (MGI) | Baseline (T0) to Month 6 (T3)
  The Modified Gingival Index (MGI) is a non-invasive visual index that evaluates gingival inflammation based on changes in color, consistency, and swelling of the marginal tissues. Scores range from 0 (normal, healthy gingiva) to 4 (severe inflammation with spontaneous bleeding). It does not require probing. The mean score per patient is used to assess the effectiveness of treatment.
Change in interproximal plaque accumulation measured by Approximal Plaque Index (API) | Baseline (T0) to Month 6 (T3)
  The Approximal Plaque Index (API) quantifies dental plaque located on interproximal surfaces. After applying a disclosing agent, the presence or absence of plaque is visually evaluated on approximal areas. The score is calculated as the percentage of plaque-positive sites over the total number of interproximal sites examined. Lower values indicate better interproximal hygiene.
Change in global plaque distribution measured by Plaque Control Record (PCR%) | Baseline (T0) to Month 6 (T3)
  The Plaque Control Record (PCR%) provides an overview of plaque presence across all four surfaces (buccal, lingual, mesial, distal) of each tooth. After staining with a plaque disclosing agent, the number of plaque-positive surfaces is recorded and divided by the total number of surfaces examined, expressed as a percentage. This index is used to monitor the effectiveness of plaque control strategies.
Change in localized gingival inflammation measured by Papillary-Marginal-Gingival Index (PMGI) | Baseline (T0) to Month 6 (T3)
  The Papillary-Marginal-Gingival Index (PMGI) assesses inflammation specifically in the interdental papilla and marginal gingiva through visual inspection. Scores range from 0 (normal appearance) to 5 (severe inflammation with ulceration and spontaneous bleeding). This score allows detection of early localized inflammatory changes not always reflected in broader indices.
Change in soft tissue loss measured by Gingival Recession (R) | Baseline (T0) to Month 6 (T3)
  Gingival Recession (R) is defined as the apical migration of the gingival margin with respect to the cementoenamel junction (CEJ), measured in millimeters. It reflects soft tissue loss and root exposure. Clinical measurements are used to monitor whether the intervention prevents further recession or contributes to soft tissue stabilization.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.